CLINICAL TRIAL: NCT01250301
Title: Complementing Current NHS Stop Smoking Service Treatments for Smokers With Behavioural Replacement: The Role of De-nicotinised Cigarettes
Brief Title: De-nicotinised Cigarettes Study
Acronym: Denic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Hayden McRobbie, Dr. Hayden McRobbie, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: qmul200910
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: Smoking Cessation; Tobacco Dependence; De-nicotinised cigarettes
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- De-nicotinised cigarettes + standard treatment (Experimental)
  Interventions: Other: De-nicotinised cigarettes + standard treatment
- Standard treatment (Active Comparator)
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: De-nicotinised cigarettes + standard treatment — Participants will receive de-nicotinised cigarettes to use as required for 2 weeks after their quit day. These cigarettes are intended to provide a replacement for the behavioural and sensory aspects of smoking without supplying nicotine.
  Participants will also receive standard NHS Stop Smoking Service treatment. This is a combination of weekly behavioural support and medication (e.g. nicotine replacement therapy/varenicline).
  Other Names: NHS Stop Smoking Service; De-nicotinised cigarettes
  Arms: De-nicotinised cigarettes + standard treatment
Other: Standard Treatment — Participants will receive standard treatment from the NHS Stop Smoking Service.
  Arms: Standard treatment

SUMMARY:
The aim of this study is to determine if using a behavioural replacement for smoking (de-nicotinised cigarettes; DNCs), in addition to standard treatment during the first two weeks after the target quit date, can reduce urges to smoke over the first 4-weeks of abstinence. Two hundred smokers who want to quit will be recruited from the community. They would all receive standard smoking cessation treatment from the NHS Stop Smoking Service (NHS SSS), which uses a combination of stop smoking medication (e.g. nicotine replacement therapy, Champix) and motivational support. On their target quit date, participants would be randomised to receive behavioural replacement ( i.e. use of de-nicotinised cigarettes) plus standard treatment for the first two weeks of their quit attempt, or to continue with standard treatment alone. De-nicotinised cigarettes are similar to standard cigarettes except that they do not deliver nicotine to the smoker. Participants will rate their urges to smoke at each week. Standard NHS SSS measures will also be taken in addition to user acceptability ratings and reactions to smoking cues.

The hypothesis is that complementing current NHS SSS treatments with de-nicotinised cigarettes, to address the non-nicotine factors associated with smoking and to help extinguish smoking behaviour, would result in lower urges to smoke than standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* Seeking treatment to stop smoking

Exclusion Criteria:

* Pregnant or breastfeeding
* Acute psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Urges to smoke in first week of abstinence | 1 week
  Differences in urges to smoke in the first week of abstinence between participants who receive a behavioural replacement (DNCs) plus standard NHS SSS treatment, with those who receive standard NHS SSS treatment alone, will be measured by the Mood and Physical Symptoms Scale (MPSS; West & Hajek, 2004).

SECONDARY OUTCOMES:
Change in ratings of tobacco withdrawal symptoms, measured by the MPSS | First 4 weeks of abstinence (from baseline- 4 weeks post-quit)
CO-validated continuous abstinence rates | 4-weeks
  CO-validated continuous abstinence rates will be measured 1-4 weeks following the target quit day in the standard treatment condition and 1-4 weeks following cessation of DNCs in the DNC condition.
Acceptability and user reactions to DNCs | 2 weeks
Urges to smoke 24 hours after quitting, measured by the MPSS | 24 hours
Profile of adverse effects up to 12 weeks post quitting | 12 weeks
Reactions to smoking cues | 12 weeks
  The differences in reactions to smoking cues between the 2 groups will be measured with smoking-related images and by the Cue Exposure Subscale of the Wisconsin Inventory for Smoking Dependence (WISDM-68; Piper, et al., 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Hayden McRobbie, Principal Investigator — Queen Mary University of London
Locations (1):
- Tobacco Dependence Research Unit, London, United Kingdom